CLINICAL TRIAL: NCT05103865
Title: Animal-Assisted Therapy in the Residential Treatment of Schizophrenia and Addictions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miguel Monfort Montolio (Other)
Responsible Party: Sponsor-Investigator, Miguel Monfort Montolio, Sponsor-investigator, Cardenal Herrera University
Organization: Cardenal Herrera University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAT S&A
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Diagnosis, Dual (Psychiatry)
Keywords: Animal-assisted therapy; everyday life skills; schizophrenia; residential treatment; dual pathology
MeSH Terms: conditions — Disease; Schizophrenia | interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (EG) (Experimental)
  Interventions: Behavioral: Animal-assisted therapy (AAT)
- Control group (Active Comparator)
  Interventions: Other: usual treatment

INTERVENTIONS:
Behavioral: Animal-assisted therapy (AAT)
  Other Names: ATT
  Arms: Experimental group (EG)
Other: usual treatment
  Arms: Control group

SUMMARY:
Animal-assisted therapy (AAT) is a complementary intervention of therapy that has shown positive results in the treatment of various pathologies. This study assesses the viability of the implementation and the efectiveness of an AAT program in patients diagnosed with substance abuse disorder and associated mental disorders (dual pathology).

DETAILED DESCRIPTION:
Animal assisted therapy (AAT) is a complementary intervention to therapy that presents positive results in the treatment of different pathologies. The study assesses the implementation and effectiveness of a TAA program in patients diagnosed with substance use disorder and schizophrenia spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-5 criteria for substance abuse disorder and the presence of schizophrenia
* Voluntary participant in the study and having signed the informed consent

Exclusion Criteria:

* Patients whose functioning could be altered by factors not specifically related to addictive pathology or mental disorder (severe cognitive impairment, intellectual deficiency or language barrier)
* Animal-specific phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
The Life Skills Profile questionnaire (LSP) | Change from Life Skills at 3-6-9 months (12 minutes)
  This questionnaire evaluates aspects of functioning that affect daily activities and the adaptation of people with mental illnesses in the community. It contains 39 items that are grouped into self-care, social-interpersonal behaviour, communication-social contact, non-personal social behaviour and autonomous life
Barrat impulsiveness scale (BIS-11) | Change from impulsiveness at 3-6-9 months (12 minutes)
  This instrument is composed of 30 items distributed into three sub-scales: nonplanning, motor and attentional. The total impulsiveness score was also obtained.
Calgary Depresión Scale for Schizophrenia (CDSS) | Change from Depresión at 3-6-9 months (12 minutes)
  El cuestionario es un intrumento estructurado, adminisitrado por un clínico de forma heteroaplicada para población adulta, con un tiempo aproximado de administración de entre 10 y 30 minutos, y aborada el área terapéutica relativa a la sintomatología de los trastornos depresivos.
Rosenberg Self-Esteem Scale | Change from self.-esteem at 3-6-9 months (12 minutes)
  The questionnaire consists of 10 statements of the feelings that the person has about himself. Five of the statements are addressed positively (items 1, 2, 4, 6 and 7) and 5 negatively (items 3, 5, 8, 9 and 10).
Positive and negative symptom scale (PANSS) | Change from Positive and negative symptom at 3-6-9 months (12 minutes)
  It is a semi-structured and hetero-applied questionnaire for the adult population. The application time is between 30-60 minutes and evaluates the positive and negative symptoms of schizophrenia and other psychotic disorders.